CLINICAL TRIAL: NCT04565535
Title: "Effect of Novel Donor Lifestyle Optimisation Protocol on Liver Regeneration in Live Liver Donors: a Randomised Control Pilot Study"
Brief Title: Effect of Novel Donor Lifestyle Optimisation Protocol on Liver Regeneration in Live Liver Donors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ILBS-LIVEDONORS-02
Record Dates: First submitted 2020-09-02; First posted 2020-09-25 (Actual); Last update posted 2023-05-30 (Actual); Status verified 2023-05

CONDITIONS: Liver Regeneration

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Experimental): Liver donors undergoing lifestyle optimisation
  Interventions: Behavioral: Novel donor lifestyle optimisation protocol
- Control arm (No Intervention): Liver donors who continue normal lifestyle.

INTERVENTIONS:
Behavioral: Novel donor lifestyle optimisation protocol — Diet based on calorie requirement as calculated by indirect calorimetry. Daily exercise.
  Arms: Intervention arm

SUMMARY:
Steatosis in case of live liver donors is on the rise and around 20- 40 % of prospective liver donors are estimated to have hepatic steatosis. Significant steatosis has been shown to be associated with inferior donor outcomes after liver transplant. Dietary and lifestyle modification has been shown to reduce steatosis and may help improve the donor outcomes after liver transplant. Donors will be randomized between two groups; one will be put under donor lifestyle optimization protocol and the other shall follow normal diet and lifestyle. Donors under optimization protocol would undergo diet modification in the form of healthy, low fat, high protein diet along with exercise for 2 weeks prior to the expected date of surgery. Investigations including liver volumetric assessment, LFT's , lipid profile , Fibroscan shall be done prior to initiation of the diet and then following completion of the 2 weeks of lifestyle modification before surgery. The intraoperative parameters including intraoperative blood loss shall be assessed and a liver biopsy will be taken intraoperatively to assess for steatosis and liver regeneration markers including CK7 and Ki 67 will be assessed. Following surgery, the liver regeneration in donor shall be assessed by doing a liver volumetry by Computed Tomography (CT) at POD7. Post surgery, the donor shall undergo daily LFT's, PT-INR and the time to its normalization and serum bilirubin shall be assessed. Markers of liver regeneration shall also be assessed initially a day before surgery and then at POD 1, 3 and 7.

DETAILED DESCRIPTION:
All prospective donors provisionally planned for donor hepatectomy excluding those undergoing left lateral hepatectomy will be informed regarding the current study and informed written consent will be taken from donors willing to participate in the study. After step II evaluation of the donors, they will be randomized into two groups. First group will be put under donor lifestyle optimization protocol and the other shall follow normal diet and lifestyle. Donors under optimization protocol would undergo diet modification in the form of healthy, low fat, high protein diet along with exercise for 2 weeks prior to the expected date of surgery. If the expected date of surgery is delayed because of any cause, the proposed lifestyle optimization shall continue till the date of surgery. Step I of the evaluation including Blood group, coagulation profile, LFT, KFT, Viral serology, Liver attenuation index on Non contrast CT scan of abdomen and a Fibroscan shall be done. After step I investigations are found to be normal, patient would be subjected to step II evaluation consisting of CECT abdomen with liver volumetry including total liver volume, right lobe volume without MHV using ,expected remnant volume using software for analysis of CT volumes, MRCP for biliary anatomy, TFT and lipid profile. Body composition analysis, Fibroscan, lipid profile and LFT shall be done prior to initiation of the diet and then following completion of the 2 weeks of lifestyle modification. The intraoperative parameters including intraoperative blood loss shall be assessed. Intra operative liver biopsy will be taken from segment IV after completion of hepatectomy from all the donors undergoing donor hepatectomy using a core needle biopsy(B Braun® 18g). Precautions will be taken to take adequate tissue samples and avoid subcapsular sampling. Hemostasis of the needle tract will be obtained by use of electro thermal energy source. The core liver biopsy will be sent in formalin containing bottle to the histopathologist. Liver biopsy will be done independently by two expert histopathologists. Any abnormal histopathological finding will be noted, degree of steatosis assessed and regenerative markers from the tissue including CK7 and Ki67 will be assessed. Following surgery, the liver regeneration in donor shall be assessed by doing a liver volumetry at POD7 and POD 14. Following donor hepatectomy, routine parameters like LFT, PT-INR will be documented and the post operative day of normalisation of PT-INR and Serum Bilirubin will be noted. The volumetry of the regenerated liver will be done at day 7 and day 14 in all the donors. Seum level of liver regenerative markers shall(including HGF, IL6, TNF alpha, TGF beta, INF alpha) will be assessed on a day before surgery and then at Post operative day 1, 3 and 7. Liver function tests and PT-INR would be evaluated daily for one week. . In the post operative period , any surgical complication arising will be assessed till first month after surgery and the donor outcomes will be monitored. Complications shall be assessed based on Clavien Dindo Classification.

On follow ups liver function tests will be performed weekly for 1 month and then at monthly intervals till 3 months after surgery. At this time, any long term complication will be assessed.

Study population: Donors undergoing donor hepatectomy after giving informed written consent to be a part of the study.

Study Design: Randomised Control Pilot Study

Study Period: From time of ethical clearance to October 2021.

Sample Size: All the donors planned for donor hepatectomy meeting the inclusion criteria from time of clearance from ethical committee to october 2021 will be enrolled in this study following which randomization will be done on basis of computer generated numbers. Anticipated sample size would be 30 in each group after exclusion.

Inclusion Criteria

All donors planned for donor hepatectomy and found fit in step II evaluation.

Those who give consent to be a part of the study.

Exclusion criteria Patients refusing to consent for the study

Donor of ALF patients.

Donors undergoing left lateral hepatectomy.

Donors found unfit after step I/II evaluation.

Intervention: Diet and lifestyle modification group will receive customized two week diet plan which would consist of calorie restricted(based on basal requirement calculated by Harris Benedict Equation), high protein(25%), low fat(15%) diet along with regular exercise (brisk walk for 45 min/day). Assessment of compliance will be checked by calling each donor twice every week and during their regular weekly follow ups as well.

ELIGIBILITY:
Inclusion Criteria:

* All donors planned for donor hepatectomy and found fit in step II evaluation.

Those who give consent to be a part of the study.

Exclusion Criteria:

* Patients refusing to consent for the study

Donor of ALF patients.

Donors undergoing left lateral hepatectomy.

Donors found unfit after step I/II evaluation.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
To study difference in Liver regeneration in Live Liver Donors on basis of: Post operative day of normalization of serum bilirubin and PT-INR between both the groups. | post operative day 1 - day 14
  Serum Bilirubin and PT-INR levels will be measured and their times of normalisation will be taken as markers for regeneration of liver.
Percentage growth of liver(on basis of CT Volumetry) | post operative day 7 and post operative day 14
  liver volumetry will be don eat POst operative day 7 and 14 to assess the percentage growth of liver by doing a CT volumetry.

SECONDARY OUTCOMES:
To study difference in Steatosis in both groups on basis of intra operative liver biopsy. | Intra operative.
  Steatosis on basis of intra operative core needle liver biopsy will be seen by the pathologist by histopathological assessment of the core needle biopsy specimen.
To study difference in Serum level of markers of liver regeneration after liver transplant in both the groups. | Pre op day 14 to post op day 7
  Blood Markers of liver regeneration including Hepatocyte growth factor(HGF), Interleukin 6(IL6), TNF alpha, TGF beta, INF alpha will be assessed.
To study difference in Rates of early graft dysfunction in recipients in both the groups. | Day 1-14
  daily liver function tests and Pt-INR will be done in case of recipients and their levels seen to report the number of recipients having early graft dysfunction.
To study difference in Body composition analysis and fibroscan before and after lifestyle modification. | at the time of enrollment to pre operative day( 2 weeks).
  Changes in body composition analysis using Bioelectrical impedance analysis and fibroscan will be done.
To study difference in Intraoperative blood loss, post op stay in the hospital and complication rates between both the groups | post operative day 0 to post operative day 14
  Difference in intra operative blood loss, post operative stay in the hospital and the complications(as per clavien dindo classification) will be noted.

CONTACTS AND LOCATIONS:
Overall Officials: Viniyendra Pamecha, FEBS, Study Director — Institute of Liver & Biliary Sciences
Locations (1):
- Institute of Liver & Biliary Sciences, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Barth RJ Jr, Mills JB, Suriawinata AA, Putra J, Tosteson TD, Axelrod D, Freeman R, Whalen GF, LaFemina J, Tarczewski SM, Kinlaw WB. Short-term Preoperative Diet Decreases Bleeding After Partial Hepatectomy: Results From a Multi-institutional Randomized Controlled Trial. Ann Surg. 2019 Jan;269(1):48-52. doi: 10.1097/SLA.0000000000002709. PMID 29489484
- [Background] Reeves JG, Suriawinata AA, Ng DP, Holubar SD, Mills JB, Barth RJ Jr. Short-term preoperative diet modification reduces steatosis and blood loss in patients undergoing liver resection. Surgery. 2013 Nov;154(5):1031-7. doi: 10.1016/j.surg.2013.04.012. Epub 2013 Jun 27. PMID 23809869
- [Background] Cho JY, Suh KS, Lee HW, Cho EH, Yang SH, Cho YB, Yi NJ, Kim MA, Jang JJ, Lee KU. Hepatic steatosis is associated with intrahepatic cholestasis and transient hyperbilirubinemia during regeneration after living donor liver transplantation. Transpl Int. 2006 Oct;19(10):807-13. doi: 10.1111/j.1432-2277.2006.00355.x. PMID 16961772
- [Background] Nakamuta M, Morizono S, Soejima Y, Yoshizumi T, Aishima S, Takasugi S, Yoshimitsu K, Enjoji M, Kotoh K, Taketomi A, Uchiyama H, Shimada M, Nawata H, Maehara Y. Short-term intensive treatment for donors with hepatic steatosis in living-donor liver transplantation. Transplantation. 2005 Sep 15;80(5):608-12. doi: 10.1097/01.tp.0000166009.77444.f3. PMID 16177634
- [Derived] Gupta A, Patil NS, Mohapatra N, Benjamin J, Thapar S, Kumar A, Rastogi A, Pamecha V. Lifestyle Optimization Leads to Superior Liver Regeneration in Live Liver Donors and Decreases Early Allograft Dysfunction in Recipients: A Randomized Control Trial. Ann Surg. 2023 Sep 1;278(3):e430-e439. doi: 10.1097/SLA.0000000000005836. Epub 2023 Mar 13. PMID 36912445